CLINICAL TRIAL: NCT03765567
Title: Placement of Antibiotic Powder in Wounds During the Emergency Room (POWDER) Study
Brief Title: Placement of Antibiotic Powder in Wounds During the Emergency Room
Acronym: POWDER
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: United States Army Institute of Surgical Research (U.S. Federal Agency); San Antonio Military Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSC20180520H; W81XWH-18-2-0074 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2018-12-04; First posted 2018-12-05 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Open Fracture
Keywords: infection; vancomycin; topical antibiotic; antibiotic prophylaxis
MeSH Terms: conditions — Fractures, Open; Infections | interventions — Vancomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Intervention Arm (Experimental): Subjects randomized to the Intervention Arm will receive usual care plus two (2) grams of Vancomycin powder administered topically. In the emergency room prior to surgical intervention, a qualified member of the study team or clinical team member will apply 2 grams of vancomycin powder directly to the open fracture site such that all visible surfaces of the wound are completely and uniformly covered, including bone edges.
  Interventions: Drug: Vancomycin
- Control Arm (No Intervention): Subjects randomized to the Control Arm will receive usual care for open long bone fracture as determined by the treating physician.
- Observational Arm (No Intervention): Subjects who otherwise meet the criteria to be included in the study but are not able to provide consent, either themselves or through a Legally Authorized Representative, will be placed in the Observational Arm and receive usual care with no experimental intervention.

INTERVENTIONS:
Drug: Vancomycin — 2 vials of Vancomycin 1g powder will be applied topically to the open fracture wound site.
  Other Names: NDC (National Drug Code) 67457-340-01; Topical vancomycin; Vancomycin powder
  Arms: Intervention Arm

SUMMARY:
This is the first prospective controlled study to determine whether the topical application of vancomycin powder reduces infection-related complications when applied to open fracture injuries in the acute emergency department setting.

DETAILED DESCRIPTION:
Open fracture injuries are highly susceptible to infection and infection-related complications. The current routine treatment for these injuries includes the use of systemic IV antibiotics. However, open fracture injuries often have compromised blood supply, reducing the amount of antibiotic that reaches the target tissue while increasing risk of injury to non-target organs. This trial aims to evaluate the effectiveness of early application of a topical vancomycin antibiotic powder on open fracture wounds, in combination with the usual treatment, in reducing the risk of infection seen in these injuries.

ELIGIBILITY:
Inclusion Criteria:

* Subject or Legal Authorized Representative (LAR) is willing and able to provide written informed consent.
* Adult 18 years of age or older.
* Open fracture of the humerus, radius, ulna, femur, tibia, and/or fibula.
* 24 hours or less has elapsed from the estimated time of injury to study intervention.

Exclusion Criteria:

* Time from injury > 24 hours.
* Subjects who have received acute operative care (e.g., washout in the operating room or fixation) of the open fracture at an outside facility.
* Subject or LAR speaks neither English nor Spanish. Note that subjects that are unable to participate in the consent process (e.g. intoxication, poly-trauma, will be enrolled into the observational arm where passive data collection will occur).
* High-potency antibiotic powder or solution applied to the wound prior to enrollment. Simple ointment (i.e., bacitracin ointment) or antibiotic-impregnated dressings will be permitted.
* Documented allergies or serious reactions to vancomycin. History of uncomplicated "red man syndrome" will not be considered a reason for exclusion.
* Pregnant subjects. If the subject is a female of childbearing potential, and she states that she is likely to be pregnant, a pregnancy test will be performed; if negative, the subject will be eligible for enrollment.
* Prisoners.
* Participation in other clinical research involving investigational antimicrobial products within 30 days of randomization.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-10-05 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Deep-space infection rate at prophylaxis site | Within one year of injury date
  The percentage of participants who develop an infection of the study open fracture requiring post-operative surgical intervention within one year of injury.

SECONDARY OUTCOMES:
Superficial infection rate requiring post-operative medical intervention | Within one year of injury date
  The percentage of participants who develop an infection of the study open fracture that requires post-operative medical intervention, including addition or change of antibiotic, bedside application of incision & drainage, needle aspiration, and bedside application of a drain.
Unplanned repeat visit rate | Within one year of injury date
  The percentage of participants who experience an unscheduled medical encounter related to open fracture-site infection.
Readmission rate for open fracture infection | Within one year of injury date
  The percentage of participants who are readmitted to the hospital due to infection or complication of the study open fracture. Included in this assessment is sepsis and sepsis-related conditions arising from an open fracture infection.
Death rate | Within one year of injury date
  The rate of death among participants from presumed or documented open fracture site infection, determined by documentation through reliable diagnostic means.

CONTACTS AND LOCATIONS:
Overall Officials: Robert A De Lorenzo, MD, Principal Investigator — University of Texas
Locations (2):
- United States (2):
  - University Hospital, San Antonio, Texas
  - San Antonio Military Medical Center, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared through the use of the REDCap Web-based distributed data collection system. All sharing of data will conform to currently established DOD HRPO (Department of Defense Human Research Protection Office) human subject protection practices and will be in compliance with all appropriate state and federal confidentiality requirements and privacy guidelines.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be made available within one year of study completion.
Access Criteria: Research data obtained through this study will be made available to researchers and/or the general public as requested. The limitations on this policy are that data will not generally be available until such a time that it is submitted for publication. While data will be provided in a timely fashion, the actual timelines of availability of requested data will be specific to the data requested and any special sensitivity of the requested data set.